CLINICAL TRIAL: NCT05423431
Title: Clinical Protocol for the Retrospective Evaluation of a Commercially Available Hydrogel Spacer
Brief Title: Retrospective Evaluation of a Commercially Available Hydrogel Spacer (BP-009)
Status: Completed | Type: Observational
Sponsor: BioProtect (Industry)
Responsible Party: Sponsor
Other Study IDs: BP-009
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Prostate; Prostate Cancer; Spacer; Perirectal spacer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radiation with Hydrogel Spacer: Males at least 18 years of age, who underwent radiation therapy with a hydrogel spacer in place.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Assessment of rectal dosimetry change from pre-insertion to post-insertion in subjects with prostate cancer who have undergone radiotherapy with a hydrogel spacer.

SUMMARY:
Dosimetry efficacy of the hydrogel spacer.

DETAILED DESCRIPTION:
Single arm study for evaluation of dosimetry following use of a commercially available hydrogel spacer implanted in up to 20 males who underwent radiotherapy treatment for prostate cancer. Study utilized pre and post gel insertion CT images to determine endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Males
* At least 18 years of age
* Undergone external beam or brachy radiation therapy with a hydrogel spacer in place

Exclusion Criteria:

* Clinical and pathological data are not available
* Invasive adenocarcinoma that is extracapsular and demonstrates posterior extension

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Prostate Cancer
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Dosimetry Changes | 1 Month
  Assessment of rectal radiation exposure as compared between rectal dose volume histograms calculated for pre and post hydrogel injection

SECONDARY OUTCOMES:
Prostate to rectum spacing | 1 Month
  Prostate to rectum spacing as measured post hydrogel insertion based on CT simulation scans done after hydrogel insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Radiation Centers of New York ("ARC"), Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No